CLINICAL TRIAL: NCT00961714
Title: Evaluation of Safety and Effectiveness of the OsseoFix™ Spinal Fracture Reduction System in Treating Spinal Compression Fracture
Brief Title: OsseoFix™ Spinal Fracture Reduction System in Treating Spinal Compression Fracture
Acronym: OsseoFix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrew study
Sponsor: Alphatec Spine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-02-A
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Vertebral Compression Fractures
Keywords: VCF

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OsseoFix (Experimental): Osseofix is an titanium expandable device similar to a vascular stent that is placed in the fractured vertebral body to provide a structure in which bone cement (polymethylmethacrylate) is inserted. It is intended to be used in the thoracolumbar spine between levels T6 through L5.
  Interventions: Device: OsseoFix Spinal Fracture Reduction System

INTERVENTIONS:
Device: OsseoFix Spinal Fracture Reduction System — All enrolled into the study will be receiving the OsseoFix if meet inclusion / exclusion criteria.

SUMMARY:
The OsseoFix Spinal Fracture Reduction System facilitates the treatment of spinal fractures by providing internal fixation and stabilization using a titanium implant in conjunction with OsseoFix+™ polymethylmethacrylate (PMMA) bone cement.

The purpose of the study is to provide reasonable assurance on safety and effectiveness of the OsseoFix Spinal Fracture Reduction System for market release approval in the US.

This investigational device is intended to restore biomechanical integrity to a vertebral body that has suffered a painful compression fracture in the thoracic or lumbar spine between levels T6 and L5.

DETAILED DESCRIPTION:
This is a prospective, multi-center clinical study designed to evaluate safety and effectiveness of the OsseoFix Spinal Fracture Reduction System used with PMMA bone cement relative to the clinical expectations for treatment of vertebral compression fractures (VCFs). The study will be conducted at up to 15 investigational centers in the United States in 115 (up to 125) subjects with one or two vertebral compression fractures between levels T6 and L5 implanted with the investigational device(s).

Baseline screening will be completed to determine eligible subjects. VCFs will be confirmed by magnetic resonance imaging (MRI), or by a CT / bone scan. These diagnostic tests will be utilized to confirm that there are no retropulsed bone fragments. Subjects who meet all inclusion criteria and do not have any exclusion criteria will be scheduled to receive the OsseoFix Spinal Fracture Reduction System.

Subjects that are enrolled will be implanted with the OsseoFix Spinal Fracture Reduction System through a postero-lateral approach to the anterior vertebral body using instruments specifically designed for this procedure.

Radiographs will be taken at each follow-up visit, including baseline and post-operatively. Subject's perception of pain will be assessed using the Visual Analogue Scale (VAS). Functional outcomes will be measured using the Oswestry Disability Index (ODI) and Short Form- 36 (SF-36) questionnaires as well as their neurologic status. The VAS, ODI, SF-36 and neurologic status will be measured at baseline, 4-week, 3-month, 6-month and 12-month follow-up visits. Overall patient-satisfaction will be evaluated at all post-implant scheduled follow-up visits. Adverse event will be the recorded in all scheduled and non-scheduled visits.

The endpoint analysis will be performed and submitted when all implanted subjects have completed their 12-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 5o years of age.
* Legal US citizen with ability to read and write.
* Acute painful fracture (≤2 months) between T6 to L5 as evidenced by plain radiography, CT / Bone scan, and/or magnetic resonance imaging.
* Subject is...

  * Non-Standard Treatment:

    * Inability to tolerate prolonged conservative care due to intractable pain (VAS 70/100) with maximum tolerated medication for at least 2 weeks, but less than 6 weeks; OR
    * Inability to tolerate prolonged immobilization due to other comorbid conditions aggravated by immobility for at least 2 weeks, but less than 6 weeks; OR
    * Intolerance of or adverse reaction to available pain medications for at least 2 weeks, but less than 6 weeks; OR
    * Hospitalization secondary to pain for at least 2 weeks, but less than 6 weeks.
  * Standard Treatment:

    * Has undergone at least 6 weeks of conservative care.
* Have a self assessment VAS score ≥ 50 mm at the Baseline visit.
* Have 30% or greater disability score on ODI at the Baseline visit.
* Anterior wedge deformity with no less than 5% and no more than 75% loss of anterior cortical height as compared to the posterior cortical height of the same vertebral body.
* Bone mineral density (BMD) T-score of -1.5 or less, as determined by a DEXA scan.
* Intact posterior cortical vertebral body wall.
* Type A compression fractures according to AO classification of spinal vertebral fractures.
* If a transpedicular approach is utilized the pedicle diameter must be equal to or greater than 6.5 mm; however, if an extrapedicular approach is utilized there is not a minimum pedicle width requirement.
* Subject is willing and able to provide informed consent and agrees to release medical information for purposes of this study (HIPAA authorization) and to return for scheduled follow-up evaluations.

Exclusion Criteria:

* Significant vertebral collapse defined as more than 75% of original vertebral height or less than 5% or a burst or pedicle fracture with posterior cortical wall disruption.
* Presence of healed fracture at the intended treatment level(s) based on a CT / bone scan or MRI.
* Compression fractures requiring treatment at 3 or more levels.
* Spinal/Foraminal canal compromised.
* Significant deformity/instability indicated by:

  * Segmental kyphosis > 30 degrees, or
  * translation > 4 mm.
* VAS back pain score of < 50 mm.
* ODI score of < 30%.
* Have a documented active systemic or local infection, such as AIDS, hepatitis, with a WBC greater than 11.5 and a temperature greater than 101.5°F.
* Spinal surgery in the thoracic and/or lumbar region within the past year
* Previous kyphoplasty or vertebroplasty at involved level or level above or below treated level.
* Spinal arthrodesis within 2 adjacent levels of fracture.
* Non-ambulatory prior to fracture.
* Greater than Grade 1 spondylolisthesis at level of fracture.
* Scoliosis > 10 degrees.
* BMI > 40.
* Severe cardiopulmonary deficiencies.
* Pregnant.
* Type I or II diabetes without controlled A1C level.
* Achondrogenesis disorders.
* Active malignancy, hemangiomas at the operative level(s), or multiple myeloma.
* No generally accepted medical contraindication to spinal surgery and/or general anesthesia, such as coagulopathy with a threshold for INR at 1.5 or less, and platelet count 100,000.
* A life expectancy less than the study duration or undergoing palliative care.
* Trauma injuries aside from vertebral compression fracture(s).
* Injuries that violate the posterior vertebral cortex and/or posterior column.
* Active litigation.
* Currently on workman's compensation.
* Autoimmune disorders.
* Non-spine pain that requires daily Opioids.
* Systemic long-term steroid use - greater than 6 months.
* Active multiple sclerosis or neurologic deficit caudal to fracture.
* Currently an alcohol, solvent, or drug abuser.
* Psychiatric or cognitive impairment that, in the opinion of the investigator, would interfere with the subject's ability to comply with the study requirements.
* History of allergies to any of the device components including but not limited to commercially pure titanium, titanium alloy, polymethylmethacrylate or Zirconium Oxide (ZrO2)
* Incarcerated.
* Are currently participating in another investigational study.
* Having had another device implanted in the thoracic and/or lumbar area that would interfere with the surgical approach, study device, or follow-up evaluations.

Ages: 50 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Yue, MD, Principal Investigator — Yale University; Daniel Bennett, MD, Principal Investigator — Integrative Treatment Centers
Locations (11):
- United States (11):
  - Scripps, La Jolla, California
  - Boulder Neurosurgery Associates, Boulder, Colorado
  - South Denver Neurosurgery, Littleton, Colorado
  - Lyerly Neurosurgery, Jacksonville, Florida
  - Southwestern Orthopedic Center, Savannah, Georgia
  - SIU Phyysicians and Surgeons Division of Orthopaedics and Rehabilitation, Springfield, Illinois
  - Jewish Hospital for Advanced Medicine, Louisville, Kentucky
  - Clinical Radiology of Oklahoma, Edmond, Oklahoma
  - NeuroSpine Institute, LLC, Eugene, Oregon
  - Orthopaedic Associates of the Greater Lehigh Valley Easton Hospital, Easton, Pennsylvania
  - Neurospine Solutions, PC, Bristol, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OsseoFix
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | OsseoFix
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 15
BMI [Mean (Standard Deviation); unit: lb/in^2] | 23.7 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Back Pain Improvement at 12 Months
Description: Back pain improvement is defined as a reduction in VAS score of ≥ 20mm at 12 months from baseline
Time Frame: 12 months
Measure: Number; unit: Percentage of available participants
Arm/Group | OsseoFix
Number analyzed (Participants) | 13
Percentage of available participants | 85

2. Primary Outcome: Percentage of Participants With Functional Disability Improvement at 12 Months
Description: Functional disability improvement is defined as a reduction in ODI score by ≥ 15 points at 12 months from baseline.
Time Frame: 12 months
Measure: Number; unit: Percentage of available participants
Arm/Group | OsseoFix
Number analyzed (Participants) | 13
Percentage of available participants | 84.6

3. Primary Outcome: Absence of Device Related Subsequent Interventions or Re-treatment at the Study Treated Levels
Time Frame: 12 months
Measure: Number; unit: Percentage of participants
Arm/Group | OsseoFix
Number analyzed (Participants) | 13
Percentage of participants | 84.6

4. Secondary Outcome: Change in Pain at 12 Months as Presented by VAS, When Compared to Baseline
Description: Pain measurements determined by Visual Analog Scale (VAS) on a 100mm scale with, 0=no pain at all, to 100=worse possible pain.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OsseoFix
Number analyzed (Participants) | 13
units on a scale | -50.7 (27.2)

5. Secondary Outcome: Functional Disability Change at 12months From Baseline as Determined by ODI
Description: Improvement in functional disability as determined by ODI on a scale of 0-50, with 0=no disability at all to 50=complete disability
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OsseoFix
Number analyzed (Participants) | 13
units on a scale | -39.9 (16.8)

6. Secondary Outcome: Any Cement Extravasation Before Discharge
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | OsseoFix
Number analyzed (Participants) | 15
participants | 1

ADVERSE EVENTS:
Arm/Group | OsseoFix
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OsseoFix (N=15)
Obstructive Hydrocephalus (Nervous system disorders) | 1
Pyelonephritis (Renal and urinary disorders) | 1
Weakness (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OsseoFix (N=15)
Cardiac Arrest (Cardiac disorders) | 1
Compression Fracture (Musculoskeletal and connective tissue disorders) | 1
Elbow Abrasion (Musculoskeletal and connective tissue disorders) | 1
Fall (General disorders) | 1
Left Trochanter Bursitis (Musculoskeletal and connective tissue disorders) | 1
Nausea (Metabolism and nutrition disorders) | 1
Pain (Nervous system disorders) | 2
Rib Fracture (Musculoskeletal and connective tissue disorders) | 2
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Thoracis Abscess (Cardiac disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No